CLINICAL TRIAL: NCT03175094
Title: PLUS PINK: HHRP+ Adaptation for Women With HIV Under Community Supervision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1407014291; K23DA033858 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: HIV
Keywords: women; HIV prevention; criminal justice
MeSH Terms: interventions — Seroconversion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holistic Health Recovery Program for HIV+ Intervention (Experimental)
  Interventions: Behavioral: Holistic Health Recovery Program for HIV+
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Holistic Health Recovery Program for HIV+ — Holistic Health Recovery Program for HIV+ (HHRP+) is a CDC-recommended, evidence based behavioral (psychoeducational) group intervention focused on harm reduction principles. The investigators systematically adapted HHRP+ using findings from qualitative interviews with the target population of adult women living with and at-risk for HIV who are justice-involved (on probation, parole, or recently released from prison or jail).
  Arms: Holistic Health Recovery Program for HIV+ Intervention

SUMMARY:
After enrollment, participants will be randomized to either receive the intervention (treatment) from trained health educators or undergo observation as usual (control group). Randomization will be stratified by HIV serostatus. A control group is appropriate because participants will still receive services offered through probation and will be offered the intervention after completion of the trial. Subjects will be paid, not for participating in the intervention, but for providing research assessments. The newly adapted intervention will be delivered over no more than a 3-month period (it will be shorter if the adaptation process is supportive). Baseline assessments will assess the pre-intervention period. The 3-month assessment will be the end-of-intervention effects and the post-intervention assessments will be at 6, 9 and 12 months. HIV prevention knowledge will be assessed based on quizzes used previously for HHRP+; though final quiz content will depend on final selected materials for the intervention. Subjects will be followed for 12 months with assessments by trained research assistants.

DETAILED DESCRIPTION:
The aim of this study is to adapt and pilot test the Holistic Health Recovery Program for women with and at risk for HIV (HHRP+), a CDC evidence-based secondary HIV prevention intervention, that will serve as a framework to optimize HIV treatment outcomes and reduce HIV-associated risk for women under correctional community supervision.

Hypotheses

1. It will be feasible to recruit and retain HIV+ and at-risk women under community correctional supervision in the pilot study.
2. Using the ADAPT-ITT methods, we will be able to adequately adapt HHRP+ for HIV-infected and at-risk women under community supervision.
3. The adapted intervention will be feasible to implement and acceptable to participants.
4. The adapted intervention will produce higher measureable preliminary effects on HIV-focused treatment outcomes in the intervention group compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* female
* have laboratory confirmed HIV OR are at-risk for HIV (ever injected drugs, ever engaged in commercial sex work, were incarcerated in prison or jail within the past 2 years, had condomless sex with an HIV+ partner or partner whose HIV status is unknown in the past 90 days, or had a diagnosed sexually transmitted infection in the past 90 days),
* and are under or anticipating transfer to probation.are either a) sentenced to probation or on intensive pretrial supervision by a probation officer; b) sentenced to parole; or c) incarcerated in jail or prison in the prior 60 days.

Potential participants will be excluded

Exclusion Criteria:

* unable or unwilling to provide informed consent,
* have <3 months of remaining scheduled supervision term,
* or are threatening to staff

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Change in HIV knowledge from baseline | 3 months
  HIV knowledge quiz with scores ranging from 0-100, a higher score indicating better knowledge

SECONDARY OUTCOMES:
Change in Sex-related risk behaviors over time | baseline, 6 months, 12 months
  NIDA Risk Behavior Assessment (0-18 with higher scores indicating higher risk)
Change in Injection-related risk behaviors over time | baseline, 6 months, 12 months
  NIDA Risk Behavior Assessment (0-18 with higher scores indicating higher risk)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Meyer, M.D., M.S., Principal Investigator — Yale University
Locations (1):
- Yale AIDS Program, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No